CLINICAL TRIAL: NCT00575016
Title: Safety and Efficacy Study of Botulinum Toxin Type A for the Treatment of Neurogenic Overactive Bladder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated early due to enrollment challenges.
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 191622-518
Record Dates: First submitted 2007-12-13; First posted 2007-12-17 (Estimated); Results first posted 2011-10-17 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-09

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Saline Solution; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- 1 (Experimental): botulinum toxin Type A (50U); botulinum toxin Type A (200U)
  Interventions: Biological: botulinum toxin Type A (50U); botulinum toxin Type A (200U)
- 2 (Experimental): botulinum toxin Type A (100U); botulinum toxin Type A (200U)
  Interventions: Biological: botulinum toxin Type A (100U); botulinum toxin Type A (200U)
- 3 (Experimental): botulinum toxin Type A (200U)
  Interventions: Biological: botulinum toxin Type A (200U)
- 4 (Other): placebo; botulinum toxin Type A (200U)
  Interventions: Biological: Normal saline (Placebo); botulinum toxin Type A (200U)

INTERVENTIONS:
Biological: Normal saline (Placebo); botulinum toxin Type A (200U) — Placebo injection on Day 1 and botulinum toxin Type A injection 200 U > Week 12; injection into the detrusor
  Other Names: BOTOX®
  Arms: 4
Biological: botulinum toxin Type A (50U); botulinum toxin Type A (200U) — botulinum toxin Type A 50 U on Day 1 followed by botulinum toxin Type A 200 U > 12 weeks; injections into the detrusor
  Other Names: BOTOX®
  Arms: 1
Biological: botulinum toxin Type A (100U); botulinum toxin Type A (200U) — botulinum toxin Type A 100 U on Day 1 followed by botulinum toxin Type A 200 U > 12 weeks; injections into the detrusor
  Other Names: BOTOX®
  Arms: 2
Biological: botulinum toxin Type A (200U) — botulinum toxin Type A 200 U on Day 1 followed by botulinum toxin Type A 200 U > 12 weeks; injections into the detrusor
  Other Names: BOTOX®
  Arms: 3

SUMMARY:
The purpose of this study is to explore the effectiveness and safety of several doses of botulinum toxin type A in treating overactive bladder in patients with spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* Urinary incontinence as a result of neurogenic overactive bladder due to spinal cord injury
* Inadequate response to anticholinergic medication used to treat overactive bladder

Exclusion Criteria:

* History or evidence of pelvic or urologic abnormality
* Previous or current diagnosis of bladder or prostate cancer
* Urinary tract infection at time of enrollment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2007-12; Primary Completion 2010-02 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (6):
- Cairo, Egypt
- Thessaloniki, Greece
- Ahmadābād, India
- Beirut, Lebanon
- Belgrade, Serbia
- Ankara, Turkey (Türkiye)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 74 patients enrolled into the study, 73 patients received study medication and are included in the analyses. One patient was enrolled but did not receive study medication.
Groups:
- Botulinum Toxin Type A (200U): botulinum toxin Type A (200U)
- Botulinum Toxin Type A (100U): botulinum toxin Type A (100U)
- Botulinum Toxin Type A (50U): botulinum toxin Type A (50U)
- Placebo: Normal saline (placebo)
Period: Treatment Cycle 1
Arm/Group | Botulinum Toxin Type A (200U) | Botulinum Toxin Type A (100U) | Botulinum Toxin Type A (50U) | Placebo
Started | 17 | 21 | 19 | 17 (1 pt randomized to Placebo never received treatment)
Completed | 8 (3 pts from 200U group entered Cycle 2) | 16 (11 pts from 100U group entered Cycle 2) | 15 (8 pts from 50U group entered Cycle 2) | 12 (9 pts from Placebo group entered Cycle 2)
Not Completed | 9 | 5 | 4 | 5
Period: Treatment Cycle 2
Arm/Group | Botulinum Toxin Type A (200U) | Botulinum Toxin Type A (100U) | Botulinum Toxin Type A (50U) | Placebo
Started | 31 (All patients received 200U in Treatment Cycle 2.) | 0 (All patients received 200U in Treatment Cycle 2.) | 0 (All patients received 200U in Treatment Cycle 2.) | 0 (All patients received 200U in Treatment Cycle 2.)
Completed | 30 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Botulinum Toxin Type A (200U) | Botulinum Toxin Type A (100U) | Botulinum Toxin Type A (50U) | Placebo | Total
Number analyzed (Participants) | 17 | 21 | 19 | 17 | 74
Age, Customized [Number; unit: participants]
  < 40 years | 13 | 13 | 16 | 11 | 53
  Between 40 and 64 years | 4 | 8 | 3 | 6 | 21
  Between 65 and 74 years | 0 | 0 | 0 | 0 | 0
  >= 75 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 2 | 1 | 10
  Male | 14 | 17 | 17 | 16 | 64

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Number of Weekly Episodes of Urinary Incontinence
Description: Change from baseline in the weekly frequency of incontinence episodes at Week 6 after the first treatment. Incontinence is defined as involuntary loss of urine as recorded in a patient bladder diary. A negative number change from baseline indicates a reduction in incontinence episodes (improvement).
Time Frame: Baseline, Week 6
Population: Modified Intent-To-Treat: defined as all patients who were randomized (started study) and received treatment
Measure: Mean (Standard Deviation); unit: Number of Weekly Episodes
Arm/Group | Botulinum Toxin Type A (200U) | Botulinum Toxin Type A (100U) | Botulinum Toxin Type A (50U) | Placebo
Number analyzed (Participants) | 17 | 21 | 19 | 16
Number of Weekly Episodes
  Baseline | 28.8 (20.26) | 37.8 (27.63) | 26.3 (19.29) | 24.6 (9.08)
  Week 6 | -15.8 (18.01) | -14.1 (23.90) | -7.7 (11.52) | -8.6 (8.12)

2. Secondary Outcome: Change From Baseline in Maximum Cystometric Capacity (MCC)
Description: Change from baseline in MCC at week 6. MCC represents the maximum volume of urine the bladder holds. A positive number change from baseline represents an improvement (increase) in maximum volume of urine the bladder holds.
Time Frame: Baseline, Week 6
Population: Modified Intent-To-Treat: defined as all patients who were randomized (started study) and received treatment
Measure: Mean (Standard Deviation); unit: Milliliters (mL) of urine
Arm/Group | Botulinum Toxin Type A (200U) | Botulinum Toxin Type A (100U) | Botulinum Toxin Type A (50U) | Placebo
Number analyzed (Participants) | 17 | 21 | 19 | 16
Milliliters (mL) of urine
  Baseline | 214.2 (96.56) | 161.6 (66.13) | 213.9 (135.41) | 189.8 (103.56)
  Week 6 | 183.7 (197.63) | 220.1 (183.05) | 136.8 (189.37) | 117.4 (173.51)

3. Secondary Outcome: Change From Baseline in Maximum Detrusor Pressure (MDP)
Description: Change from baseline in MDP during first involuntary detrusor contraction at week 6. MDP represents the maximum pressure (peak amplitude) in the bladder during the first involuntary contraction of the bladder muscle. The greater the negative number change from baseline, the better the improvement.
Time Frame: Baseline, Week 6
Population: Modified Intent-To-Treat: defined as all patients who were randomized (started study) and received treatment
Measure: Mean (Standard Deviation); unit: Centimeters of water (cm H2O)
Arm/Group | Botulinum Toxin Type A (200U) | Botulinum Toxin Type A (100U) | Botulinum Toxin Type A (50U) | Placebo
Number analyzed (Participants) | 17 | 21 | 19 | 16
Centimeters of water (cm H2O)
  Baseline | 62.9 (72.05) | 54.2 (41.47) | 52.7 (39.51) | 45.9 (36.82)
  Week 6 | -33.0 (58.06) | -29.4 (39.67) | -20.1 (22.07) | -2.1 (27.65)

ADVERSE EVENTS:
Description: The safety population was used to calculate the number of participants at risk for SAEs and AEs and is the total number of patients that were randomized AND treated. S(AE)s are displayed for the placebo-controlled treatment Cycle 1.
Arm/Group | Botulinum Toxin Type A (200U) | Botulinum Toxin Type A (100U) | Botulinum Toxin Type A (50U) | Placebo
Serious Adverse Events (participants affected / at risk) | 2/17 | 2/21 | 2/19 | 6/16
Other Adverse Events (participants affected / at risk) | 11/17 | 17/21 | 11/19 | 13/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Botulinum Toxin Type A (200U) (N=17) | Botulinum Toxin Type A (100U) (N=21) | Botulinum Toxin Type A (50U) (N=19) | Placebo (N=16)
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Sudden death (General disorders) | 1 | 1 | 0 | 0 — Both events not related to study medication.
Malaria (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Intestinal stoma (Surgical and medical procedures) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Botulinum Toxin Type A (200U) (N=17) | Botulinum Toxin Type A (100U) (N=21) | Botulinum Toxin Type A (50U) (N=19) | Placebo (N=16)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Hyperchlorhydria (Gastrointestinal disorders) | 1 | 2 | 1 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Anal inflammation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 2 | 0 | 3
Asthenia (General disorders) | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 1 | 0
Sudden death (General disorders) | 1 | 1 | 0 | 0 — Both events not related to study drug
Urinary tract infection (Infections and infestations) | 7 | 11 | 7 | 10
Malaria (Infections and infestations) | 0 | 0 | 0 | 1
Orchitis (Infections and infestations) | 0 | 0 | 0 | 1
Acute tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Infected skin ulcer (Infections and infestations) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 2
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
White blood cells urine positive (Investigations) | 0 | 0 | 0 | 1
Red blood cells urine positive (Investigations) | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1
Panic disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 2 | 1 | 5
Haematuria (Renal and urinary disorders) | 1 | 0 | 2 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Vesical fistula (Renal and urinary disorders) | 1 | 0 | 0 | 0
Epididymitis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Intestinal stoma (Surgical and medical procedures) | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Due to recruitment difficulties, study enrollment was stopped early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less